CLINICAL TRIAL: NCT00242021
Title: Fatty Acid Composition of a Fat Supplement on Energy Intake, Satiety and Fat Metabolism in Lean and Obese Men
Brief Title: The Effect of Fatty Acid Composition on Energy Intake and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Ministry of Health, Welfare and Sport (Unknown)
Responsible Party: Dr. W.J. Pasman, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P6468
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity
Keywords: Satiety, ad libitum food intake, fatty acids, hormones
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Fatty acid composition of a margarine (spread)

SUMMARY:
The objective of the study is to investigate the effect of fatty acid composition of a fat supplement:

1. acutely (after single intake) on subjective and objective measurements of hunger, satiety and wellness, on energy intake, and postprandial hormonal changes;
2. in the long-term (after one week) on (regulators of) fat tissue metabolism.

DETAILED DESCRIPTION:
One of the physiological factors regulating the food intake pattern is satiety. Satiety is defined as the absence of ingestive motivation, which ends when the next meal is initiated (Blundell et al., 1996). Food intake affects a number of physiological objective parameters in blood known to be involved in signaling satiety, such as glucose (Melanson et al, 1999; Chapman et al, 1999; Campfield et al, 1996), insulin (Speechly et al, 2000) and cholecystokinin (CCK) (Gutzwiller et al., 2000; Beglinger et al., 2001; French et al., 2000; Degen et al., 2001; Burton-Freemanet al., 2002, 2004). More recently, the gastric hormone ghrelin was identified as a marker for hunger and meal initiation (De Graaf et al, 2004). Ghrelin concentrations in blood were highly correlated with subjective measures of appetite. PYY, a gut hormone produced postprandially, will be measured in this study because it has been mentioned that this hormone inhibits food intake (Batterham et al., 2003). The baseline level of PYY is lower in obese subjects than in lean subjects. The two groups different in body weight will therefore show different baseline levels, and perhaps different curves as well.

Humans do not only eat in response to a metabolic or physiological need. Humans also respond to a significant extend to other internal subjective and emotional signals (cues). The exact relations between the physiological internal signals and subjective and emotional internal signals are not known. Besides also external and social factors modulate physiological-derived hunger and satiety signals.

In the present clinical trial, the effect of fatty acid composition of a fat supplement will be studied on hunger and satiety. In the supplement a mixture of fatty acids known for their satiating effect will be tested and will be compared with a control supplement containing fatty acids normally consumed with breakfast.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the health and lifestyle questionnaire, physical examination and results of the pre-study laboratory tests;
2. Males aged between 18 - 60 years at Day 01 of the study;
3. Normal weight subjects and overweight/obese subjects, Body Mass Index (BMI) will be at least two units different between the heaviest normal weight and the lightest overweight subject, the largest contrast between groups will be aimed at, e.g normal weight BMI between 18 and 25 kg/m2 and overweight/obese BMI between 27.5-35 kg/m2;
4. Regular Dutch eating habits as assessed by P6468 F02 and used to breakfast consumption;
5. Non restrained eater, defined as a score of < 2.5 in lean and <3.25 in obese men on the Dutch Eating Behaviour Questionnaire;
6. Appropriate veins for blood sampling/cannula insertion according to TNO;
7. Voluntary participation;
8. Having given written informed consent;
9. Willing to comply with the study procedures;
10. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years;
11. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study;
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances;
3. Having a history of medical or surgical events that may significantly affect the study outcome, including any psychiatric history, and metabolic or endocrine disease, or any gastro-intestinal disorder or hypertension;
4. Use of medication that may influence appetite, and/or sensory functioning within 14 days before day 01, except paracetamol;
5. Allergic reaction to chlorhexidine and/or lidocaine (anaesthetic solution);
6. Having a history of or current alcohol consumption of more than 28 units/week;
7. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening;
8. Mental or physical status that is incompatible with the proper conduct of the study;
9. Reported chronic and/or excessive mental or physical strain;
10. Reported slimming or medically prescribed diet;
11. Reported vegan, vegetarian or macrobiotic;
12. Use food supplement(s) and not willing to stop intake after the medical screening;
13. Smoking;
14. Claustrophobia;
15. Practicing heavy physical exercise > 5 hours/week;
16. Recent blood donation (<1 month prior to the start of the study) and not willing to give up blood donation during the study;
17. Personnel of TNO Quality of Life, their partner and their first and second degree relatives;
18. Not having a general practitioner;
19. Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Subjective and objective measurements of hunger, satiety and wellness, on energy intake, and postprandial hormonal changes

SECONDARY OUTCOMES:
After one week supplementation the effect on (regulators of) fat tissue metabolism will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands